CLINICAL TRIAL: NCT01744145
Title: Early Pneumonia Intervention to Prevent Chronic Complications in Patients Age 40 and Above
Brief Title: Effect of Exercise and Education After Pneumonia
Acronym: EPICC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough enrollment
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 255021-4
Record Dates: First submitted 2012-09-20; First posted 2012-12-06 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2016-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Interventional 40-60 (Active Comparator): Interventional group aged 40-60
  Interventions: Other: Interventional 40-60
- Control 40-60 (No Intervention): Control group aged 40-60
- Interventional 60 and above (Active Comparator): Interventional group aged 60 and above
  Interventions: Other: Interventional 60 and above
- Control 60 and above (No Intervention): Control group aged 60 and above

INTERVENTIONS:
Other: Interventional 40-60 — This group will receive the intervention aged 40-60
  Arms: Interventional 40-60
Other: Interventional 60 and above — This group will receive the intervention aged 60 and above.
  Arms: Interventional 60 and above

SUMMARY:
The mortality rate and quality of life is effected in patients with pneumonia, especially in the older population.

The end point of this study is to improve quality of life by and interventional exercise and education. Patients will be randomized at admission and enrolled into the study. They will be assessed with various performance and quality of life indicators before, during and after the study, and exercise tolerance will be assessed throughout and after.

DETAILED DESCRIPTION:
The purpose of this research study is to assess improvement in functional status and quality of life of patients 40 years of age and older patients hospitalized for community acquired pneumonia and healthcare associated pneumonia with a multi-disciplinary program of exercise, education and psychological support. This study will use a randomized, controlled clinical trial design. The total number of patients enrolled will be 120, divided into two groups of 60 patients each. One group will have patients age 40 to 60 and second group will have patients age 60 and above. Stratified randomization will be done to divide these into two (control group and intervention group) equal groups with 30 patients each. The primary endpoint is improvement in quality of life indices. Secondary endpoints are improvement in functional status, change in 6 minute walk test, exercise intolerance, immunization, occult desaturation and change in body weight of patients hospitalized for community acquired pneumonia with a multi-disciplinary program of exercise, education and, psychological support. Eligibility includes age 40 and above at the time of admission, diagnosis of CAP and HCAP via radiographic and PNA symptoms, discharge to home, ability to read and sign informed consent to participate, ability to perform procedures/exercises involved in the study and ability to comprehend educational component of program.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CAP or HCAP via radiographic imaging and symptoms of pneumonia Age 40 and above.
2. Discharge to home.
3. Ability to read and sign consent.
4. Ability to perform in procedures/exercise.
5. Ability to understand educational component of the program.
6. Antibiotic administration for pneumonia within 12 hours of admission.

Exclusion Criteria:

1. Severe lung diseases like ILD(Interstitial Lung disease), ARDS (Adult Respiratory Distress Syndrome.)
2. Ventilator dependent patients.
3. Discharge to nursing home.
4. Comorbidity that could limit exercise training.
5. Dementia, Schizophrenia or any active severe psychiatric disorder.
6. Any Active Malignancy or diagnosis of Lung malignancy.
7. Inability to attend program two times per week.
8. Recent myocardial infarction within two months.
9. Unstable angina, Heart failure (NYHA class III and IV.)
10. Patients with pneumonia who did not receive antibiotics within 12 hours of admission.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
improvement in quality of life indices | one year
  patients in the interventional group will undergo exercise and education after a pneumonia infection to see if the quality of life is effected by a rehab program

SECONDARY OUTCOMES:
improvement in functional status | one year
change in 6 minute walk test | one year
exercise intolerance | one year
immunization | one year
  Patients will be assessed to see if education offered in the interventional group will effect compliance with vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Shalinee Chawla, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hosptial, Mineola, New York, United States